CLINICAL TRIAL: NCT05057676
Title: Evaluation of an Online Course Designed to Support the Adoption of Healthier Diet and Self-Care Routines in Multiple Sclerosis Patients
Brief Title: Autoimmune Intervention Mastery Course Study
Acronym: AIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Terry L. Wahls (Other)
Responsible Party: Sponsor-Investigator, Terry L. Wahls, Clinical professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202103542
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis; Clinically Isolated Syndrome; Fibromyalgia; Post Acute Sequelae of COVID-19; Cancer in Remission With Persisting Fatigue
Keywords: diet; self care
MeSH Terms: conditions — Multiple Sclerosis; Fibromyalgia; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Wait list control
Who Masked: Investigator
Masking Description: Investigator will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Autoimmune Intervention Mastery Course (AIM) online course (Experimental): This arm will begin the intervention immediately after randomization
  Interventions: Behavioral: Immediate Autoimmune Intervention Mastery Course (AIM); Behavioral: Immediate Question and Answer sessions. (AIM Q and A sessions)
- Delayed Autoimmune Intervention Mastery Course (Other): This is the control arm.
  Interventions: Behavioral: Delayed Autoimmune Intervention Mastery Course (delayed AIM course); Behavioral: Delayed AIM Question and Answer sessions

INTERVENTIONS:
Behavioral: Immediate Autoimmune Intervention Mastery Course (AIM) — Immediate access to an on line audio and video course with education about strategies to grow and improve resilience, diet quality, exercise, stress reduction and self-care
  Other Names: AIM course
  Arms: Intervention Autoimmune Intervention Mastery Course (AIM) online course
Behavioral: Immediate Question and Answer sessions. (AIM Q and A sessions) — Immediate access to videos answering common questions about the course concepts. One video released each week, 7 videos total.
  Other Names: AIM Q and A sessions
  Arms: Intervention Autoimmune Intervention Mastery Course (AIM) online course
Behavioral: Delayed Autoimmune Intervention Mastery Course (delayed AIM course) — Delayed access to an on line audio and video course with education about strategies to grow and improve resilience, diet quality, exercise, stress reduction and self-care
  Arms: Delayed Autoimmune Intervention Mastery Course
Behavioral: Delayed AIM Question and Answer sessions — Delayed access to videos answering common questions about the course concepts. One video released each week, 7 videos total.
  Other Names: Delayed AIM Q and A sessions
  Arms: Delayed Autoimmune Intervention Mastery Course

SUMMARY:
The goal of this project is to critically evaluate the effectiveness of using an online program to improve diet and self-care in patients with multiple sclerosis (MS), clinically isolated syndrome (CIS), fibromyalgia, post acute sequela of covid, and cancer in remission with persisting fatigue.

DETAILED DESCRIPTION:
The goal of this project is to critically evaluate the effectiveness of using an online program to improve diet and self-care in patients with multiple sclerosis (MS), clinically isolated syndrome (CIS), fibromyalgia, post acute sequela of covid, and cancer in remissin with persisting fatigue. The cancer patients must be patients at the University of Iowa Holden Cancer Center.

Once eligibility criteria are determined and consent is obtained, participants would work through the course modules like a non-graded online course. There are exercises and personal assessments within the course participants are asked to take to build upon each other to increase the success of the experience while taking the course.

Throughout the course there will be modules that will discuss an inner game plan, food intervention plan, physical intervention plan, and an increased resilience plan. The fourth module suggests different strategies that participants can do to improve their health beyond food and exercise. These types of things would include supplements, light therapy, detoxification, improved sleep, stress reduction, and other ways to enhance their body's resilience.

Investigators ask that participants inform and work with their healthcare team to personalize their treatment and determine if the suggested strategies mentioned in the course are appropriate for their healthcare path. This will provide dietary education to a larger sample size compared to what has been studied in the past. The study may include more patients that have limited resources, including but not limited to, money and location for access to registered dietitians with expertise in dietary instruction for patient s diagnosed with multiple sclerosis and CIS. There is interest in education and support that can be delivered via an online platform that can lead to improved diet quality and self-care routines for multiple sclerosis and autoimmune patients.

This study will use a randomized single-blind wait list control design to evaluate the impact of an online course that teaches the modified Paleolithic diet, nutrient dense vegetarian diet and Mediterranean diets, stress reduction and exercise strategies using commercially available online course for autoimmune patients. Data will be collected in the short-term (after 3 months) and long-term (at the end of 6 months ) to analyze the impact of an online wellness program QoL and related outcomes among people with CIS and MS, fibromyalgia, post acute sequela of covid, and cancer in remission wiht persisting fatigue.

The study will use a 7-day window to collect baseline assessments. Participants will use a personal email that does not contain identifying information to participate in the study. Participants will be asked to complete all baseline assessments. This email and password will be used for access to the online course materials. Patients will be randomized to the intervention arm based upon the baseline modified fatigue impact score.

Patients will receive access to the online program and 7 group support videos (released one per week or 7 weeks total). Participants will access the course materials using the study assigned email.

The proposed study will consist of virtual-only participants and will have 3 virtual visits every 3 months (months 0, 3, and 6). Online questionnaires will be sent to the participants to assess fatigue and quality of life. Dietary assessments will include a questionnaire through a web-based tool after baseline, at month 3, and month 6.

ELIGIBILITY:
Inclusion Criteria:

* self-reported multiple sclerosis
* self-reported clinically isolated syndrome

OR self-reported post-acute sequelae of COVID (PASC), also known as long COVID, with a confirmed laboratory test of COVID-19 infection, persisting fatigue and neuropsychiatric symptoms for longer than 6 months after confirmation of COVID diagnosis,

OR self-reported diagnosis of fibromyalgia as documented by their treating specialist or primary care provider,

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis 54 Quality of Life Mental Health (MS 54 QoL MH) | baseline to 3 months
  Change in (MS 54 QoL MH) survey questions mean scores, range 0-100, higher number is better.
Multiple Sclerosis 54 Quality of Life Mental Health (MS 54 QoL MH) | baseline to 6months
  Change in (MS 54 QoL MH) survey questions mean scores, range 0-100, higher number is better.
Multiple Sclerosis 54 Quality of Life Physical Health (MS 54 QoL PH) | baseline to 3 months
  Change in (MS 54 QoL PH) survey questions mean scores, range 0-100, higher number is better.
Multiple Sclerosis 54 Quality of Life Physical Health (MS 54 QoL PH) | baseline to 6 months
  Change in (MS 54 QoL PH) survey questions mean scores, range 0-100, higher number is better.
Short form 36 (SF 36) | baseline to 3 months
  Change in (SF 36) survey questions mean scores, range 0-100, higher number is better.
Short form 36 (SF 36) | baseline to 6 months
  Change in (SF 36) survey questions mean scores, range 0-100, higher number is better.
The Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-FS): | baseline to 3 months
  FACIT-FS is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function, which can be completed in less than 5 minutes.10 Each question provides 5 ordinal response options ("not at all," "a little bit," "somewhat," "quite a bit," and "very much"). Each item contributes equally (item score range=0-4) to a total score that ranges from 0 to 52, where higher scores represent less fatigue.
The Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-FS): | baseline to 6 months
  FACIT-FS is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function, which can be completed in less than 5 minutes.10 Each question provides 5 ordinal response options ("not at all," "a little bit," "somewhat," "quite a bit," and "very much"). Each item contributes equally (item score range=0-4) to a total score that ranges from 0 to 52, where higher scores represent less fatigue.

SECONDARY OUTCOMES:
Modified Fatigue Impact Scale | baseline to 3 months
  Change in MFIS survey questions, scores range from 0-84, lower score is better.
Modified Fatigue Impact Scale | baseline to 6 months
  Change in MFIS survey questions, scores range from 0-84, lower score is better.
vegetable and fruit intake | baseline to 3 months
  Change in number of servings of vegetables consumed per day, servings range from 0 to 9 or more
vegetable and fruit intake | baseline to 6 months
  Change in number of servings of vegetables consumed per day, servings range from 0 to 9 or more
added sugar intake | baseline to 3 months
  change in the grams of added sugar consumed each day, grams range from 0 to 100
added sugar intake | baseline to 6 months
  change in the grams of added sugar consumed each day, grams range from 0 to 100
calcium intake | baseline to 3 months
  change in calcium intake, range 0 to 2000 mg
calcium intake | baseline to 6 months
  change in calcium intake, range 0 to 2000 mg
Servings of whole grains consumed | baseline to 3 months
  change in number of servings of whole grains consumed, range 0 to 6 or more servings
Servings of whole grains consumed | baseline to 6 months
  change in number of servings of whole grains consumed, range 0 to 6 or more servings
Fibromyalgia Impact Questionnaire Revised | baseline to 3 months
  Pain Rating (0-10 Low to High Scale) survey questions with higher score indicating greater impact
Fibromyalgia Impact Questionnaire Revised | baseline to 6 months
  Pain Rating (0-10 Low to High Scale) survey with 15 items with higher score indicating greater impact
Brief Pain Inventory | baseline to 3 months
  Interference (0-10 Low to High Scale) 15 survey items with higher score indicating greater intensity
Brief Pain Inventory | baseline to 6 months
  Range 0-10(Low to High Scale) survey with higher score indicating greater pain intensity
FM Disease activity (FIQR) | baseline to 3 months
  0-100( Low to High Scale)21 survey items used to evaluate function, overall impact, and symptoms in patients with fibromyalgia.
FM Disease activity (FIQR) | baseline to 6 months
  0-100 (Low to High Scale)21 survey items used to evaluate function, overall impact, and symptoms in patients with fibromyalgia. High score indicating more severe symptoms.
Pain scale | baseline to 3 months
  0-10 (low to high) 13 survey items used to evaluate feelings about pain.
Pain catastrophizing scale | baseline to 6 months
  052 (low to high) 13 survey items used to evaluate feelings about pain. Higher scores indicating more severe feelings about pain related problems
Functional Assessment of Cancer Therapy - General (FACT-G) | baseline to 3 months
  measures health-related QoL covering 5 domains: physical well-being (7 items), family/social well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and fatigue-specific items (13 items).10 These items are scored on a 5-point Likert scale, where 0 = "not at all" and 5 = "very much," with a recall period over the past 7 days. Domain scores can be calculated by summing the scores for each domain, and/or a total score by summing the scores for all domains, with higher scores representing better functioning. General guidelines estimate for the FACT-G minimally important difference (MID), is 4-7 points. The total score ranges from 0-108.
Functional Assessment of Cancer Therapy - General (FACT-G) | baseline to 6 months
  measures health-related QoL covering 5 domains: physical well-being (7 items), family/social well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and fatigue-specific items (13 items).10 These items are scored on a 5-point Likert scale, where 0 = "not at all" and 5 = "very much," with a recall period over the past 7 days. Domain scores can be calculated by summing the scores for each domain, and/or a total score by summing the scores for all domains, with higher scores representing better functioning. General guidelines estimate for the FACT-G minimally important difference (MID), is 4-7 points. The total score ranges from 0-108.

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Wahls, MD, Principal Investigator — University of Iowa
Locations (1):
- Univeristy of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wahls TL, Chenard CA, Snetselaar LG. Review of Two Popular Eating Plans within the Multiple Sclerosis Community: Low Saturated Fat and Modified Paleolithic. Nutrients. 2019 Feb 7;11(2):352. doi: 10.3390/nu11020352. PMID 30736445
- [Background] Wahls T, Scott MO, Alshare Z, Rubenstein L, Darling W, Carr L, Smith K, Chenard CA, LaRocca N, Snetselaar L. Dietary approaches to treat MS-related fatigue: comparing the modified Paleolithic (Wahls Elimination) and low saturated fat (Swank) diets on perceived fatigue in persons with relapsing-remitting multiple sclerosis: study protocol for a randomized controlled trial. Trials. 2018 Jun 4;19(1):309. doi: 10.1186/s13063-018-2680-x. PMID 29866196
- [Background] Chenard CA, Rubenstein LM, Snetselaar LG, Wahls TL. Nutrient Composition Comparison between a Modified Paleolithic Diet for Multiple Sclerosis and the Recommended Healthy U.S.-Style Eating Pattern. Nutrients. 2019 Mar 1;11(3):537. doi: 10.3390/nu11030537. PMID 30832289
- [Background] Titcomb TJ, Bisht B, Moore DD 3rd, Chhonker YS, Murry DJ, Snetselaar LG, Wahls TL. Eating Pattern and Nutritional Risks among People with Multiple Sclerosis Following a Modified Paleolithic Diet. Nutrients. 2020 Jun 20;12(6):1844. doi: 10.3390/nu12061844. PMID 32575774
- [Background] Wahls TL, Titcomb TJ, Bisht B, Eyck PT, Rubenstein LM, Carr LJ, Darling WG, Hoth KF, Kamholz J, Snetselaar LG. Impact of the Swank and Wahls elimination dietary interventions on fatigue and quality of life in relapsing-remitting multiple sclerosis: The WAVES randomized parallel-arm clinical trial. Mult Scler J Exp Transl Clin. 2021 Jul 31;7(3):20552173211035399. doi: 10.1177/20552173211035399. eCollection 2021 Jul-Sep. PMID 34377527
- [Background] Lee JE, Titcomb TJ, Bisht B, Rubenstein LM, Louison R, Wahls TL. A Modified MCT-Based Ketogenic Diet Increases Plasma beta-Hydroxybutyrate but Has Less Effect on Fatigue and Quality of Life in People with Multiple Sclerosis Compared to a Modified Paleolithic Diet: A Waitlist-Controlled, Randomized Pilot Study. J Am Coll Nutr. 2021 Jan;40(1):13-25. doi: 10.1080/07315724.2020.1734988. Epub 2020 Mar 26. PMID 32213121
- [Background] Bisht B, Darling WG, Grossmann RE, Shivapour ET, Lutgendorf SK, Snetselaar LG, Hall MJ, Zimmerman MB, Wahls TL. A multimodal intervention for patients with secondary progressive multiple sclerosis: feasibility and effect on fatigue. J Altern Complement Med. 2014 May;20(5):347-55. doi: 10.1089/acm.2013.0188. Epub 2014 Jan 29. PMID 24476345
- [Background] Bisht B, Darling WG, White EC, White KA, Shivapour ET, Zimmerman MB, Wahls TL. Effects of a multimodal intervention on gait and balance of subjects with progressive multiple sclerosis: a prospective longitudinal pilot study. Degener Neurol Neuromuscul Dis. 2017 Jun 26;7:79-93. doi: 10.2147/DNND.S128872. eCollection 2017. PMID 30050380
- [Background] Irish AK, Erickson CM, Wahls TL, Snetselaar LG, Darling WG. Randomized control trial evaluation of a modified Paleolithic dietary intervention in the treatment of relapsing-remitting multiple sclerosis: a pilot study. Degener Neurol Neuromuscul Dis. 2017 Jan 4;7:1-18. doi: 10.2147/DNND.S116949. eCollection 2017. PMID 30050374
- [Derived] Titcomb TJ, Sherwood M, Ehlinger M, Saxby SM, Shemirani F, Eyck PT, Wahls TL, Snetselaar LG. Evaluation of a web-based program for the adoption of wellness behaviors to self-manage fatigue and improve quality of life among people with multiple sclerosis: A randomized waitlist-control trial. Mult Scler Relat Disord. 2023 Sep;77:104858. doi: 10.1016/j.msard.2023.104858. Epub 2023 Jun 27. PMID 37399671